CLINICAL TRIAL: NCT02976454
Title: Using a Guided Self-Help Treatment Model for Childhood Obesity Management in the Primary Care Setting
Brief Title: Guided Self-Help Obesity Treatment in the Doctor's Office - GOT Doc
Acronym: GOTDoc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kay Rhee, Associate Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R40MC29452
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Obesity
Keywords: Obesity treatment; Primary care; Guided Self-Help
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Self-Help Obesity Treatment (Experimental): Guided Self-Help obesity treatment will include 14 meetings over 6 months to mimic the structure of the proposed Medicare funding for obesity treatment for adults. These meetings will include a single one-hour meeting and 13 twenty-minute meetings that occur in the clinic. During this time, the health coach will assess patient/parent readiness to engage in behavior change, assess barriers and facilitators to behavior change, engage in behavior change and problem solving, and provide feedback and accountability.
  Interventions: Behavioral: Guided Self-Help Obesity Treatment
- Family-based behavioral obesity treatment (Active Comparator): The active control group will receive usual care, i.e. PCP provides obesity management using decision support tools in the electronic health record and refers to a tertiary care program at the academic center. This program is the traditional family-based behavioral weight control program which consists of 20 one-hour, group-based sessions over 6 months.
  Interventions: Behavioral: Family-based behavioral obesity treatment

INTERVENTIONS:
Behavioral: Guided Self-Help Obesity Treatment — Guided Self-Help obesity treatment will be provided by a health coach in the clinic. The treatment involves 14 sessions: 1 one-hour session and 13 twenty-minute sessions with the health coach who will provide behavioral obesity treatment.
  Other Names: Guided self-help
  Arms: Guided Self-Help Obesity Treatment
Behavioral: Family-based behavioral obesity treatment — Traditional family-based, group-based behavioral weight control program. The treatment involves 20 hourly group-based sessions for parents and children separately, which occurs weekly for 16 weeks, then every other week for the last 2 months (4 session).
  Other Names: FBT
  Arms: Family-based behavioral obesity treatment

SUMMARY:
One-third of our nations' children are overweight or obese (OW/OB). The cornerstone of obesity treatment involves intensive family-based behavioral therapy, yet these programs often exist in tertiary care academic settings that have long wait lists and are too far away for families to access. Primary care providers (PCP) have been called on by several organizations to be the front line of obesity management, yet they are limited by a lack of time, resources, and skills. Thus, if we are to offer effective obesity management in the healthcare setting, other care models need to be developed and tested. The goal of this proposal is to deliver Guided Self-Help (GSH) treatment of childhood obesity in the primary care setting. This program relies on classic behavioral therapy strategies, self-regulation theory, and provides the support needed for patient/family self-management of weight loss. Implementing this program in the primary care setting will increase our ability to deliver nutrition and weight-related counseling in the primary care office and serve patients closer to home, thereby increasing access to effective treatment, improving adherence to recommended changes, and meeting the goals of Healthy People 2020.

DETAILED DESCRIPTION:
Currently 1/3 of our nation's children are overweight or obese. The goal of Healthy People 2020 is to reduce the proportion of children who are obese and increase the proportion of primary care visits that include nutrition and weight-related counseling. However, there are a lack of resources and providers that can offer effective weight-related counseling and treatment. Gold-standard family-based weight control programs for children are often provided at tertiary care academic centers and can be difficult to access. Furthermore, primary care providers (PCPs), who have been identified as key players in the treatment of childhood obesity, are not well-equipped to address this issue, engage in behavior modification/lifestyle counseling, or provide effective treatment in the primary care setting. As a result, new models of care are needed so that a greater proportion of overweight/obese (OW/OB) children and their parents can access care and receive quality treatment for obesity. The investigators propose to train health coaches in the primary care setting to deliver Guided Self-Help (GSH) treatment of childhood obesity. Implementing this program in the primary care setting will increase our ability to deliver nutrition and weight-related counseling in the primary care office and serve patients closer to home, thereby increasing access to effective treatment, improving adherence to recommended changes, and meeting the goals of Healthy People 2020.

The goal of this study is to conduct a pragmatic clinical trial in two large pediatric practices in San Diego County (n=200) where 38% and 39% of children are OW/OB. The intervention group will receive GSH (14 sessions over 6 months) delivered by a health coach in the clinic. The control group will receive usual care, i.e. PCP provides obesity management using decision support tools in the electronic health record and refers to a tertiary care program (20 sessions over 6 months) at the academic center.

ELIGIBILITY:
Inclusion Criteria:

* an OW/OB child (BMI ≥ 85th%ile for age and gender) in the family who is between the ages of 5 and 13 years old
* parent who is responsible for food preparation willing to participate
* parent who can read English or Spanish at a minimum of a 5th grade level
* family who is willing to commit to attendance at all assessment visits
* family not moving out of the San Diego area within the time frame of the study.

Exclusion Criteria:

* child who is taking medications that may impact weight
* child or parent with a psychiatric or behavioral illness that will impact their ability to participate in treatment
* child with physical difficulties that limit the ability to exercise

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in BMI percentile | 6 months and 1 year
  Change in BMI percentile within and between study groups
Difference in percentage of sessions that were attended | 6 months
  Difference in percentage of sessions that were attended between groups

SECONDARY OUTCOMES:
Societal cost for each 0.1 unit BMI z-score change | 6 months and 1 year
  Cost-effectiveness from a societal perspective including cost of delivering intervention, parental costs, and primary care office costs
Activity Support scale | 6 months
  Difference in parent support behaviors to encourage physical activity between groups
Parent self-efficacy for health related behaviors scale | 6 months
  Difference in parent self-efficacy to engage in weight loss between intervention parents and control parents
Dietary History Questionnaire II | 6 months
  Changes in child dietary behavior from baseline to post treatment
Godin Physical Activity Scale | 6 months
  Changes in child physical activity level from baseline to post treatment
Dietary Support scale (modified) | 6 months
  Difference in parent support behaviors to encourage healthy dietary behaviors between groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Rhee KE, Herrera L, Strong D, Kang-Sim E, Shi Y, Boutelle KN. Guided Self-Help for Pediatric Obesity in Primary Care: A Randomized Clinical Trial. Pediatrics. 2022 Jul 1;150(1):e2021055366. doi: 10.1542/peds.2021-055366. PMID 35712916